CLINICAL TRIAL: NCT07248163
Title: A Clinical Study of the Safety and Efficacy of Universal CAR-T Cells Targeting CD19 in the Treatment of r/r B Lymphocyte Non-Hodgkin Lymphoma
Brief Title: Universal CAR-T Cell Therapy for NHL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bioray Laboratories (Industry)
Collaborators: Shanghai Tongji Hospital (Tongji Hospital of Tongji University) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-BRL-301-02-IIT
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Non-hodgkin Lymphoma,B Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): 5×10^6/kgBW
  Interventions: Drug: BRL-301

INTERVENTIONS:
Drug: BRL-301 — The administered dose is 5×10^6/kg
  Other Names: Allogeneic Chimeric Antigen Receptor T-Cell Injection Targeting the CD19 Gene

SUMMARY:
This is a single-center, single-arm, open-label clinical study, and the sample size is set to 3-6 subjects.

DETAILED DESCRIPTION:
This is a single-center, single-arm, open-label clinical study, and the sample size is set to 3-6 subjects. Evaluating the safety, tolerability, and efficacy of BRL-301 at a dose level of 5E6/kg.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to participate in this clinical study and sign an informed consent form;
2. Age ≥ 18 years old;
3. Estimated survival time ≥ 3 months;
4. At least one measurable lesion;
5. CD19 positively expressed;
6. ECOG score 0-1；
7. Hematology, coagulation and biochemistry parameters meeting the requirements;
8. LVEF ≥ 55%;
9. No severe pulmonary disorders;

Exclusion Criteria:

1. Pregnant or lactating women;
2. Subjects who previously received allogeneic cell therapies, including allogeneic stem cell transplant;
3. Subjects who previously received anti-CD19 targeted therapy;
4. Prior treatment with any CAR-T cell product or other genetically modified T cell therapies;
5. History of Richter's transformation of chronic lymphocytic leukemia (CLL);
6. Presence of uncontrollable fungal, bacterial, viral, or other infections requiring systemic therapy;
7. Subjects with positive hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) and peripheral blood HBV DNA titer higher than the upper limit of detection; hepatitis C virus (HCV) antibody positive and peripheral blood HCV RNA positive; human immunodeficiency virus (HIV) antibody positive; syphilis test positive;
8. Severe mental disorders; history of CNS disorders (e.g., epileptic seizure, cerebrovascular ischemia/hemorrhage, dementia, cerebellar diseases, or any CNS-involved autoimmune disorders);
9. Active autoimmune disorders requiring immunotherapy, including but not limited to end organ damages caused by autoimmune disorders (e.g., Crohn's disease, rheumatoid arthritis, and systemic lupus erythematosus) in the past 2 years, or requiring systemic application of immunosuppressive drugs or other drugs for systemic control of diseases;
10. Primary immunodeficiency;
11. History of other malignancies;
12. Patients with severe cardiovascular disorders;
13. Any circumstances that possibly increase the risk of subjects or interfere with the study results as judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2027-08-15 (Estimated); Study Completion 2028-03-11 (Estimated)

PRIMARY OUTCOMES:
DLT | Within 28 Days After BRL-301 Infusion
  The number and severity of dose-limiting toxicity (DLT) events

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghi Tongji Hospital (Tongji Hospital of Tongji University), Shanghai, China

IPD SHARING:
Plan to Share IPD: No